CLINICAL TRIAL: NCT05873998
Title: Analysis of CO2/Volume and CO2-pressure Curves to Detect the Lung's Closing Pressure in Ventilated Patients
Brief Title: Detecting Lung's Closing Pressure by Capnography
Status: Completed | Type: Observational
Sponsor: Hospital Privado de Comunidad de Mar del Plata (Other)
Responsible Party: Sponsor
Other Study IDs: CP2023
Record Dates: First submitted 2023-02-28; First posted 2023-05-24 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Atelectasis
Keywords: carbon dioxide; mechanical ventilation
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adults anesthetized patients undergoing mediastinoscopy: Determination of the lung's closing pressure by pressure-CO2 and volume-CO2 curves using a slow pressure-volume curve after anesthesia induction. Later on, a standard lung recruitment maneuver followed by a positive end-expiratory pressure trial was done to detect the lung's closing pressure.
  Interventions: Diagnostic Test: Slow pressure-volume curve

INTERVENTIONS:
Diagnostic Test: Slow pressure-volume curve — Patients will be sequentially subjected to a slow pressure-volume curve and a lung recruitment maneuver
  Other Names: Lung recruitment maneuver

SUMMARY:
General anesthesia is associated with loss of pulmonary functional residual capacity and the consequent development of atelectasis and closure of the small airway.

Mechanical ventilation in a lung with reduced functional residual capacity and atelectasis increased the dynamic alveolar stress-strain, inducing a local inflammatory response in atelectatic lung areas known as ventilatory-induced lung injury. This phenomenon may appear even in healthy patients undergoing general anesthesia and predisposes them to hypoxemic episodes that can persist in the early postoperative period.

Lung recruitment maneuvers restore the functional residual capacity and, therefore, protect the lungs from lung injury. A key issue in this kind of treatment is detecting the lung's closing pressure in order to maintain the end-expiratory pressure above such a limit.

DETAILED DESCRIPTION:
This is a prospective and observational study designed to measure the lung's closing pressure. The investigators will study 20 mechanically ventilated patients scheduled for mediastinoscopy surgery under general anesthesia.

Lung mechanics and capnography will be assessed during surgery. A slow pressure-volume curve will be automatically performed by the ventilator, and the small airway closing pressure will be determined as the inflection point in the alveolar slope of the pressure-CO2 and volume-CO2 curves. Then, a lung recruitment maneuver will be applied following a descending positive end-expiratory pressure trial to determine the lung's closing pressure. The investigator will see if the lung's closing pressure found with these two techniques is similar.

ELIGIBILITY:
Inclusion Criteria:

* Age > 17 years ole
* Programmed surgery

Exclusion Criteria:

* Pregnancy
* No programmed surgery
* Hemodynamic instability
* Severe COPD
* Acute respiratory infection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing general anesthesia for mediastinoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-10 (Actual)

PRIMARY OUTCOMES:
Airway pressure | 30 minutes
  Airway pressure will be measured at the airways opening and expressed in cmH2O.
Carbon dioxide | 30 minutes
  Expired carbon dioxide will be measured at the airways opening by a main-stream capnograph, expressed in mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Nora Fuentes, PhD, Study Chair — Hospital Privado de Comunidad
Locations (1):
- Hospital Privado de Comunidad, Mar del Plata, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No